CLINICAL TRIAL: NCT03686423
Title: Reversing Diabetic Peripheral Neuropathy Through Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-00527
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Peripheral Neuropathy; Diabetes
Keywords: Exercise
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetes Mellitus; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Type 2 Diabetes and Clinical Symptoms of DPN (Experimental): Patients will be individually prescribed to a 10-week exercise program with both aerobic and resistance components. Prior to beginning the intervention, patients will participate in a maximal graded exercise test (VO2R) using a cycle ergometer with a metabolic cart and integrated ECG.
  Interventions: Procedure: Exercise Program

INTERVENTIONS:
Procedure: Exercise Program — The exercise program will combine moderate intensity aerobic exercise with lower-extremity specific resistance training. A moderate level of intensity will be calculated based on results from a maximal graded exercise test (VO2R) conducted prior to the intervention.

SUMMARY:
This project proposes a longitudinal design that uses multinuclear-MRI to evaluate the mechanistic effects of exercise on skeletal muscle function and peripheral nerve integrity in patients with diabetic peripheral neuropathy (DPN), and to determine whether exercise can reverse DPN symptoms. The investigators will prescribe a 10-week exercise program to 40 DPN patients. The investigators will acquire multinuclear-MRI data before and after the intervention that can provide mechanistic insight into the adaptations in lower leg muscle function and peripheral nerve integrity of patients with DPN, and their role in improving DPN symptoms following physical exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 40 and 70
* Clinical diagnosis of Type 2 diabetes
* Clinical diagnosis of DPN
* Have a BMI less than 40 kg/m2 (due to magnet bore restrictions)
* Able to walk unassisted

Exclusion Criteria:

* Serious cardiac pathology or musculoskeletal problems that would limit exercise ability
* MNSI score < 1
* Current open wound or history of plantar ulcer for the last 3 months
* Partial foot amputations
* Inability to ambulate without assistive device
* Stroke or other central nervous system pathology
* Stage 2 hypertension (resting blood pressure >160 systolic or >100 diastolic)
* Contraindications to 3T whole body MRI scanners (e.g., pacemaker, cerebral aneurysm clip, cochlear implant, presence of shrapnel in strategic locations, metal in the eye, claustrophobia, or other problems).
* Subjects with alcoholism, chronic drug use, chronic gastrointestinal disease, or renal or hepatic impairment
* Pregnant women and children

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Brown, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Started | 44
Completed | 29
Not Completed | 15
Not completed — Withdrawal by Subject | 9
Not completed — lost to follow up (study interrupted by COVID) | 6

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 14
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI)
Description: The BMI calculation divides an adult's weight in kilograms by their height in meters squared.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 29
kg/m^2 | 30.7 (4.2)

2. Primary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: The BMI calculation divides an adult's weight in kilograms by their height in meters squared.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 29
kg/m^2 | 30.2 (4.1)

3. Primary Outcome: Glycosylated Hemoglobin (HbA1c)
Description: The glycosylated hemoglobin test shows what a person's average blood glucose level was for the 2 to 3 months before the test. Measured via patient blood samples.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage (%) of HbA1c
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 25
percentage (%) of HbA1c | 7.4 (1.2)

4. Primary Outcome: Glycosylated Hemoglobin (HbA1c)
Description: as for outcome 3
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: percentage (%) of HbA1c
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 25
percentage (%) of HbA1c | 7.3 (1.2)

5. Primary Outcome: C-Reactive Protein Levels
Description: Measured via patient blood samples.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 25
mg/L | 4.5 (3.8)

6. Primary Outcome: C-Reactive Protein Levels
Description: Measured via patient blood samples.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 25
mg/L | 4.6 (4.5)

7. Primary Outcome: Michigan Neuropathy Screening Instrument (MNSI) Symptom Questionnaire
Description: 15-question assessment of symptoms. Responses of "yes" to items 1-3, 5-6, 8-9, 11-12, 14-15 are each counted as one point. A "no" response on items 7 and 13 counts as 1 point. Item 4 is a measure of impaired circulation and item 10 is a measure of general asthenia; neither are included in scoring. The total score ranges from 0-13; lower scores indicate less prevalent symptoms; a decrease in scores indicates symptoms decreased during the observational period.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 27
score on a scale | 5.7 (1.9)

8. Primary Outcome: Michigan Neuropathy Screening Instrument (MNSI) Symptom Questionnaire
Description: as for outcome 7
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 27
score on a scale | 4.8 (2.2)

9. Primary Outcome: MNSI Physical Exam Score
Description: Completed by physician. Assessment of abnormalities in the appearance of the feet, vibration sense, reflexes, and monofilament sensation. The total score ranges from 0-10; lower scores indicate greater physical health; a decrease in scores indicates physical health increased during the observational period.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 27
score on a scale | 3.3 (1.3)

10. Primary Outcome: MNSI Physical Exam Score
Description: as for outcome 9
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 27
score on a scale | 3.2 (1.7)

11. Primary Outcome: Calf Muscle Performance
Description: Performance will be quantified as peak ankle plantarflexion torque at 60 degrees/sec.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: newton-meters
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 26
newton-meters | 35 (15)

12. Primary Outcome: Calf Muscle Performance
Description: Performance will be quantified as peak ankle plantarflexion torque at 60 degrees/sec.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: newton-meters
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 26
newton-meters | 44 (19)

13. Primary Outcome: Physical Performance Test (PP) Score
Description: 9-item assessment of Physical Performance. The total score ranges from 0 to 36; higher scores indicate greater levels of physical performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 29
score on a scale | 31.5 (3.5)

14. Primary Outcome: Physical Performance Test (PP) Score
Description: as for outcome 13
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 29
score on a scale | 33.1 (2.7)

15. Primary Outcome: PCr Resynthesis Rate in the Gastrocnemius Muscle Groups
Description: Measured using multinuclear-MRI following a 90-second plantar flexion exercise during which resistance is applied at approximately 40% of the individual's maximum voluntary contraction. The value reported in the data table represents the average flexion across both calf muscles.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mM/seconds
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 15
mM/seconds | 35.4 (21.8)

16. Primary Outcome: PCr Resynthesis Rate in the Gastrocnemius Muscle Groups
Description: as for outcome 15
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: mM/seconds
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 15
mM/seconds | 32.3 (21.7)

17. Primary Outcome: Intramuscular Adipose Tissue (IMAT) Levels in the Gastrocnemius Muscle Groups
Description: Measured using IDEAL-MRI. IMAT levels are quantified as a percentage of total tissue in the gastrocnemius muscle groups of both calf muscles combined.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of tissue
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 28
percentage of tissue | 9.1 (4.5)

18. Primary Outcome: Intramuscular Adipose Tissue (IMAT) Levels in the Gastrocnemius Muscle Groups
Description: as for outcome 17
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: percentage of tissue
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 28
percentage of tissue | 9 (4.5)

19. Primary Outcome: IMAT Levels in the Soleus Muscle Groups
Description: Measured using IDEAL-MRI. IMAT levels are quantified as a percentage of total tissue in the soleus muscle groups of both calf muscles combined.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of tissue
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 28
percentage of tissue | 9.8 (4.1)

20. Primary Outcome: IMAT Levels in the Soleus Muscle Groups
Description: as for outcome 19
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: percentage of tissue
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 28
percentage of tissue | 9.9 (4.2)

21. Primary Outcome: Fractional Anisotropy (FA) in the Tibial Nerve
Description: FA is a scalar value between zero and one that describes the degree of anisotropy of a diffusion process. A value of zero means that diffusion is isotropic, i.e. it is unrestricted (or equally restricted) in all directions. A value of one means that diffusion occurs only along one axis and is fully restricted along all other directions. Measured using Diffusion Tensor Imaging (DTI).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 17
score on a scale | 0.32 (0.07)

22. Primary Outcome: Fractional Anisotropy (FA) in the Tibial Nerve
Description: as for outcome 21
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 17
score on a scale | 0.33 (0.05)

23. Primary Outcome: Apparent Diffusion Coefficient (ADC) in the Tibial Nerve
Description: ADC is a measure of the magnitude of diffusion (of water molecules) within tissue. Measured using DTI.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: x10^3 mm^2/s
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 17
x10^3 mm^2/s | 1.76 (0.2)

24. Primary Outcome: Apparent Diffusion Coefficient (ADC) in the Tibial Nerve
Description: ADC is a measure of the magnitude of diffusion (of water molecules) within tissue. Measured using DTI.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: x10^3 mm^2/s
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
Number analyzed (Participants) | 17
x10^3 mm^2/s | 1.81 (0.19)

ADVERSE EVENTS:
Time Frame: 10 Weeks
Arm/Group | Patients With Type 2 Diabetes and Clinical Symptoms of DPN
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 5/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Type 2 Diabetes and Clinical Symptoms of DPN (N=44)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Knee pain (Musculoskeletal and connective tissue disorders) | 1
Ventricular ectopy (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT03686423/Prot_SAP_000.pdf